CLINICAL TRIAL: NCT04525820
Title: High Dose Vitamin-D Substitution in Patients With COVID-19: a Randomized Controlled, Multi Center Study
Acronym: VitCov
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Jörg Leuppi (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Jörg Leuppi, Chief Physician, Medical University Clinic, Principal Investigator, Cantonal Hosptal, Baselland
Organization: Cantonal Hosptal, Baselland (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-01401
Record Dates: First submitted 2020-08-17; First posted 2020-08-25 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Vitamin D Deficiency; Corona Virus Infection; ARDS; Coronavirus; SARS-CoV Infection
Keywords: Covid19; Vitamin D Deficiency; ARDS; Corona Virus; High dose vitamin D
MeSH Terms: conditions — COVID-19; Vitamin D Deficiency; Coronavirus Infections; Severe Acute Respiratory Syndrome | interventions — Single Person; Vitamin D; Cholecalciferol; Therapeutics

STUDY DESIGN:
Intervention Model Description: one group receives a single high dose of vitamin D in addition to treatment as usual (TAU) the other group receives a single dose of placebo in addition to TAU
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The blinding is performed by the hospital pharmacy of the university hospital of Basel. They will provide us with packed and labeled study medication and placebo. They will provide us with medication packages for each patient which includes either high dose vitamin D and the standard medication or the placebo and the standard medication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose Vitamin D (Experimental): Patient will receive a single high dose of vitamin D (140'000) in addition to daily 800 IU of vitamin D.
  The medication be administered orally
  Interventions: Drug: Single high dose vitamin D; Drug: Treatment as usual vitamin D
- Placebo (Placebo Comparator): Patient will receive a single dose of placebo, orally administered and then treatment as usual (daily 800 IU of vitamin D, orally administered)
  Interventions: Drug: Placebo; Drug: Treatment as usual vitamin D

INTERVENTIONS:
Drug: Single high dose vitamin D — Patient receives either one dose orally of 140'000 IU (7 ml) of this drug once as an intervention treatment additionally to TAU or the patient receives 7 ml of the placebo Solution (7 ml) in addition to TAU
  Other Names: VITAMIN D3 oil 500 IU/drop
  Arms: High Dose Vitamin D
Drug: Placebo — Patient receives a single dose of a placebo solution
  Other Names: Oily placebo solution
  Arms: Placebo
Drug: Treatment as usual vitamin D — Both groups receive the treatment as usual after the single high dose or the placebo which will be 800 IU per day
  Other Names: Vitamin D3 solution 4000 IU/ml

SUMMARY:
The world is currently facing a pandemic with the coronavirus (SARS-CoV-2) which leads to the disease of COVID-19. Risk factors for a poor outcome of COVID-19 have so far been identified as older age and co-morbidity including chronic respiratory conditions such as chronic obstructive pulmonary disease (COPD) and current smoking status. Previous studies found, that vitamin D deficiency is more prevalent among patients with these risk factors. There are observational studies reporting independent associations between low serum concentrations of 25-hydroxyvitamin D (the major circulating vitamin D metabolite) and susceptibility to acute respiratory tract infection.

Vitamin D substitution in patients with COVID-19 who show a vitamin D deficiency should therefore be investigated for efficacy and safety.

The study is designed as a randomized, placebo-controlled, double blind study. The objective of the study is to test the hypothesis that patients with vitamin D deficiency suffering from COVID-19 treated under standardized conditions in hospital will recover faster when additionally treated with a single high dose of vitamin D compared to standard treatment only.

DETAILED DESCRIPTION:
The world is currently experiencing a coronavirus (SARS-CoV-2) pandemic. The disease caused by infection with this virus is known as COVID-19. Risk factors for a poor outcome of COVID-19 have so far been found to include, older age and co-morbidity including chronic respiratory conditions and current smoking status. Previous studies found, that vitamin D deficiency is more prevalent among patients with these risk factors.

There are observational studies reporting independent associations between low serum concentrations of 25-hydroxyvitamin D (the major circulating vitamin D metabolite) and susceptibility to acute respiratory tract infection. 25-hydroxyvitamin D supports induction of antimicrobial peptides in response to both viral and bacterial stimuli suggesting a potential mechanism by which vitamin D inducible protection against respiratory pathogens might be mediated. The clear functions of vitamin D in the immune system are difficult to define because the immune response is not a static process. The vitamin-D-receptor, which has also been detected in immunological cells, suggests that vitamin D can regulate some processes related to immunity. A further argument which supports a potential antiviral activity of vitamin D is the modulation of the inflammatory response. The release of pro-inflammatory cytokines by the influenza virus appeared to correlate with the severity of illness. The use of vitamin D as a prophylactic for influenza has shown promise in prevention of illness and reduction of secondary asthma in children. Inadequate vitamin D status is associated with susceptibility to upper respiratory infections in patients with chronic obstructive pulmonary disease (COPD). In the ViDiCo-trial vitamin D supplementation protected against moderate or severe exacerbation, but not upper respiratory infection, in patients with COPD. A further study retrospectively examined data from 108 patients with acute respiratory distress syndrome (ARDS) for whom a vitamin D status was available at the time of diagnosis revealed that over 95% of these patients had vitamin D deficiency. When examined according to quarterly of serum 25- hydroxyvitamin D, a consistent inverse relationship between serum 25-hydroxyvitamin D and length of hospital and ICU stay among survivors was observed. Vitamin D substitution in patients with COVID-19 who show a vitamin D deficiency should therefore be investigated for efficacy and safety.

For this purpose the investigators designed a randomized, placebo controlled double blind trial to test the hypothesis hypothesis that a single high dose of vitamin D in addition to standard treatment improves the recovery period positively in patients with COVID-19 and vitamin D deficiency compared to standard treatment only. That means, that the time of recovery is shorter in the single high dose vitamin D group relative to standard treatment group only.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Hospitalized Patient
* Ongoing COVID-19 infection
* Vitamin D deficiency defined as a serum 25-hydroxyvitamin D concentration ≤ 50nmol/l( ≤20ng/ml)
* > 18 years of age

Exclusion Criteria:

* Known hypersensitivity to one of the used products of vitamin D or indigents in the drug's composition
* Active malignancy
* Hypercalcemia
* Granulomatous disease such as sarcoidosis
* History of renal stones within the past year
* Pregnancy/breastfeeding, as evaluated through screening,
* Previous enrollment into the current study,
* Enrollment of the investigator, his/her family members, employees and other dependent persons,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Length of hospitalization | Administration to Discharge from hospital care (mean duration is between 14 and 22 days for Patients with COVID 19)
  Overall duration of the hospitalization from day of admission until the day of discharge or fatality

SECONDARY OUTCOMES:
Need of intensive care | Until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID-19)
  Did the patient need a intensive care treatment during the hospitalization (yes/no)
Lenght of the Intensive Care Treatment | Until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID-19)
  Day of admission to ICU until discharge or fatality
Overall mortality | During the length of hospitalisation (mean duration is between 14 and 22 days for Patients with COVID-19)
  Percentage of patient died during hospitalization
Development of vitamin D levels | Day 1 (Baseline) and Day 7 after the first administration of the high dose vitamin D or the placebo and at discharge (mean hospital stay is between 14 and 22 days for Patients with COVID-19)
  percentage of patients with 25-hydroxyvitamin D > 50nmol/L (>20ng/mL) at day 7
  - The values of calcium, phosphorus, 24-hydroxyvitamin D, 1.25-dihydroxyvitamin D, parathyroid hormone.
Development of sepsis | During the length of hospitalization (mean duration is between 14 and 22 days for Patients with COVID-19)
  percentage of patients developing a sepsis

OTHER OUTCOMES:
Complications due to COVID-19 | During the length of hospitalization (mean duration is between 14 and 22 days for Patients with COVID-19)
  We assess every other complications which occurs due to COVID-19
Blood pressure (BP) | Daily until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID-19)
  The BP will be assessed daily in mmHg
Heart rate | Daily until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID-19)
  The heart rate will be assessed daily in bpm
Peripheral oxygen saturation (SpO2) | Daily until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID 19)
  The SpO2 will be assessed daily in %
Percentage of patients who require oxygen | Daily until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID 19)
  Requirement for oxygen will be assessed daily (yes/no) if yes how many liters per minute
Breathing frequency | Daily until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID 19)
  Breathing frequence will be assessed daily in breaths per minute
Glasgow Coma Scale (GCS) | Daily until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID 19)
  GCS will be assessed daily 3 to 15 points. It describes the extent of impaired consciousness. 15 points means no impairment, 3 points means severe impairment of consciousness.
Percentage of patients are smokers, former smokers or lifelong non-smokers | Assessing of the smoking Status at Basleine
  Assessing the history of smoking in pack years (PY). the assessment will be made with the following options for answering Current smoker: Smoking for how many years? Cigarettes per day? Former smoker, how many years smoked? How many cigarettes per day Life-long non-smoker
Current Symptoms | Daily until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID 19)
  Assessed in No/ Mild/ Moderate /Severe
Temperature | Daily until discharge or fatality (mean duration is between 14 and 22 days for Patients with COVID 19)
  Temperature will be assessed daily in degrees celsius

CONTACTS AND LOCATIONS:
Overall Officials: Jörg D Leuppi, Professor, Study Director — Cantonal Hosptal, Baselland
Locations (2):
- Switzerland (2):
  - Cantonal Hospital Baselland Liestal, Liestal, Basel-Landschaft
  - Cantonal Hospital St. Gallen, Sankt Gallen, Canton of St. Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jaun F, Boesing M, Luthi-Corridori G, Abig K, Makhdoomi A, Bloch N, Lins C, Raess A, Grillmayr V, Haas P, Schuetz P, Gabutti L, Muser J, Leuppi-Taegtmeyer AB, Giezendanner S, Brandle M, Leuppi JD. High-dose vitamin D substitution in patients with COVID-19: study protocol for a randomized, double-blind, placebo-controlled, multi-center study-VitCov Trial. Trials. 2022 Feb 4;23(1):114. doi: 10.1186/s13063-022-06016-2. PMID 35120577